CLINICAL TRIAL: NCT02331901
Title: Cerebral Microstructural Changes Following Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Erhard Trillingsgaard Næss-Schmidt, PhD fellow, University of Aarhus
Other Study IDs: mtbi-1
Record Dates: First submitted 2014-12-23; First posted 2015-01-06 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MTBI SYMP: Mild Traumatic Brain Injury subjects with symptoms
- MTBI NO SYMP: Mild Traumatic Brain Injury subjects without symptoms

SUMMARY:
This study examine the possible microstructural changes in the middle brain after mTBI using diffusion MRI

DETAILED DESCRIPTION:
There is a need for clinical and biological markers at 2-3 month to screen people in risk of getting chronic post-concussion symptoms (PCS) but also biomarkers in the brain to find out if this group with prolonged symptoms has measurable changes in the brain which could explain the persisting symptoms.

Several biomarkers and brain areas have been investigated as possible sites of injury after mild traumatic brain injury (mTBI). The nature of the diffuse PCS makes corpus callosum (CC), thalamus (THA) and hippocampus (HIP) interesting because of their central position and connection to widespread motor, sensory and cognitive processes and other brain areas.

In most prior studies conventional magnetic resonance imaging (MRI) has failed to detect pathology especially in the later phase. Diffusional Kurtosis Imaging (DKI) and Diffusional Tensor Imaging (DTI) are more sensitive to microstructural changes and might serve as biomarkers in the middle brain after mTBI.

It is hypothesized that there will be a difference in the microstructure of the thalamus, corpus callosum and hippo campus as measured with DKI between two groups of mTBI subjects with and without PCS. Secondary it is hypothesized that DKI are more sensitive than DTI in the measure of microstructural changes.

ELIGIBILITY:
Inclusion Criteria:

* Concussion caused by a head trauma according to the diagnostic criteria recommended by the Danish Consensus Report on Commotio Cerebri within the last 2-5 months. The criteria are based recommendations by the WHO Task Force, but with the amendment, that there must have been a direct contact between the head and an object in order to rule out acceleration - deceleration traumas.
* Age 18 to 30 years at the time of the head trauma.
* Able to understand, speak and read Danish.
* Patients with symptoms at least three items on the Rivermead Post Concussion Symptoms Questionnaire (RPQ) rated as moderate or severe problem. PCS have to be subjectively rated as causing substantial impairment in daily life. Patients with out symptoms (controls) having no problems on the RPQ.

Exclusion Criteria:

* 1. Objective neurological findings from neurological examination and / or acute trauma CT scan, indicating neurological disease or brain damage.
* Previous concussion leading to persistent PCS within the last two years.
* Severe misuse of alcohol, prescription drugs and / or illegal drugs.
* Psychiatric morbidity or severe neurological disease that impedes participation in the treatment, i.e. Bipolar Disorder, autism, psychotic disorder (life time), multiple sclerosis etc..
* Suitable for MRI examination

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Mild traumatic brain injury subjects with and without symptoms 3-4 months after trauma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Diffusion kurtosis Imaging (DKI) | 2-5 month after mTBI
  MRI measurement unit

SECONDARY OUTCOMES:
Diffusion Tensor Imaging (DTI) | 2-5 month after mTBI
  MRI measurement unit

OTHER OUTCOMES:
Symptoms | 2-5 month after mTBI
  Questionnaire
Cognitive performance | 2-5 month after mTBI
  Interview and computer test

CONTACTS AND LOCATIONS:
Overall Officials: Erhard T Næss-Schmidt, PhD fellow, Principal Investigator — University of Aarhus
Locations (1):
- Region Hospital Hammel Neurocenter, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No